CLINICAL TRIAL: NCT04919278
Title: The Effects of Chiropractic on Quality of Life, Sleep and Pain in Pregnant Women
Brief Title: Ciropractic Care and Pregnant Women
Acronym: ChiroPW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barcelona College of Chiropractic (Other)
Responsible Party: Principal Investigator, Pablo Perez de la Ossa, Head of Research, Barcelona College of Chiropractic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCC2018AJ
Record Dates: First submitted 2021-06-04; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Pain, Back; Pregnancy Related; Sleep; Quality of Life
Keywords: Chiropractic
MeSH Terms: conditions — Back Pain | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will be evaluated for any health contraindication. Once reviewed they will received full spine chiropractic treatment for 4 weeks, at the rate of one adjustment per week. After three visits they will complete the outcome measures
  Interventions: Procedure: Chiropractic adjustments
- Control group (No Intervention): Paticipants will be selected amongst thse attending predelivery sessions. They receive no chiropracti care. They will complete the outcomes at the same time as the Intervention group and then 4 weeks later.

INTERVENTIONS:
Procedure: Chiropractic adjustments — Chiropractic adjustment is a procedure in which trained specialists (chiropractors) use their hands or a small instrument to apply a controlled, sudden force to a spinal joint. The goal of this procedure, also known as spinal manipulation, is to improve spinal motion and improve your body's physical function.
  Arms: Intervention group

SUMMARY:
Objective: The aim of this study is to investigate the effectiveness of Chiropractic care on pain, quality of life and sleep in pregnant women compared to a control group.

The study is designed as non-randomized controlled trial. Forty-two pregnant women at least on the 14th week of gestation will be included. Control group will include women receiving regular care, but no chiropractic care. Care will extend for 4 weeks.

Outcomes measures include sleep quality, pain and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women over the age of 18
* of at least 14 weeks gestation,
* with a good understanding of English, Spanish or French.

Exclusion Criteria:

* women over the age of 45,
* pregnancies of more than 35 weeks gestation
* high-risk pregnancies (tobacco, alcohol or substance use, diagnosed medical conditions or high blood pressure).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
SF-36 questionnaire Quality of Life | 4 weeks
  The Short Form-36 Health Survey (SF-36) is one of the most frequently used and evaluated health-related quality of life measures for pregnancy. It is composed of 36 questions (items) that evaluate both positive and negative states of health. The questionnaire assesses eight dimensions: physical functioning, role limitation from physical health problems, bodily pain, general health, vitality, social functioning, and role limitation from emotional health problems
Pittsburgh Sleep Quality Index (PSQI) | 4 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire, which evaluates sleep quality and disturbances over a period of one month. It is composed of nineteen individual items creating seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, daytime dysfunction and the total PSQI score.
Numeric pain rating scale | 4 weeks
  The Numeric Rating Scale (NRS) is among the most commonly used measures of pain intensity in clinical and research settings. The NRS is an 11-point scale, from 0 to 10 with 0 indicating "no pain" and 10 representing the "worst imaginable pain". Participants select the number that best represents their pain intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- Barcelona College of Chiropractic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No